CLINICAL TRIAL: NCT04841655
Title: Tobacco Cessation Among Smokers Under Alcohol and/or Cannabis Treatment
Acronym: ACT-ATAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Català d'Oncologia (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Althaia Xarxa Assistencial Universitària de Manresa (Other); University of Barcelona (Other); Public Health Agency of Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: PI18/01420
Record Dates: First submitted 2019-12-09; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Mental Health Disorder; Substance Abuse Drug; Alcohol Abuse; Cannabis Use; Tobacco Use; Smoking Cessation
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders; Alcoholism; Tobacco Use; Smoking Cessation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aims: To identify the predictors associated with smoking cessation in smokers under treatment for alcohol and/or cannabis treated in drug treatment centers (DTC). Methodology: Mixed methods project with qualitative and quantitative designs (three studies). Study I discussion groups: of clinical professionals of DTC to explore the barriers/facilitators of these smokers in quitting and the interventions carried out. Study II Prospective cohort of smokers in alcohol and/or cannabis treatment that will be followed-up for 12 months. Sample size: difference in incidence (exposed to cessation interventions versus non-exposed = 12 per 100 years), α = 0.05, β = 0.10, losses = 20% (n = 726). Dependent variables: self-reported and verified tobacco consumption abstinence, quit attempts, motivation, and self-efficacy. Independent variables: age, sex, the substance under treatment. Analysis: incidence, relative risk and simple and multiple logistic regression models (odds ratio and confidence interval, CI, 95%) of quitting. Study III discussion groups: with smokers under alcohol and/or cannabis treatment selected according to their typology. Analysis: of thematic content and triangulation qualitative and quantitative results. Expected results: Characterization of variables that influence tobacco cessation, to improve the design of interventions.

ELIGIBILITY:
Inclusion Criteria:

* Smokers (at least 1cig./week)
* Undertreatment for Cannabis and/or Alcohol Abuse for the first time
* >=18 years-old
* Under clinical follow-up
* Informed consent

Exclusion Criteria:

* Severe cognitive impairment
* 12-month follow-up not guaranteed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Smokers under treatment for substance abuse (alcohol and/or cannabis) from the province of Barcelona in Catalonia (Spain)
Sampling Method: Non-Probability Sample
Enrollment: 1625 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
self-reported and verified tobacco consumption abstinence | at twelve months follow-up
  self-reported and verified tobacco consumption abstinence by using CO measurement

SECONDARY OUTCOMES:
Motivation to quit | at twelve months follow-up
  self-reported and scored from a Likert scale from 0 to 10 (0= no motivation 10=high motivation)
Number of cigarettes per day | at twelve months follow-up
  self-reported
Stages of Change to quit | at twelve months follow-up
  Status of the stages of change to quit according to 5 stages proposed by Prochaska and DiClemente

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinic, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez C, Pla M, Feliu A, Enriquez M, Saura J, Cabezas C, Colom J, Suelves JM, Mondon S, Barrio P, Andreu M, Raich A, Bernabeu J, Roca X, Narvaez M, Fernandez E; Group of clinicians of the ACT_ATAC study. Clinician's perceptions and experiences with tobacco treatment in people who use cannabis: a qualitative study. Subst Abuse Treat Prev Policy. 2025 Jan 21;20(1):3. doi: 10.1186/s13011-024-00632-8. PMID 39838401
- [Derived] Feliu A, Fernandez E, Castellano Y, Enriquez M, Saura J, Cabezas C, Colom J, Suelves JM, Pla M, Parejo M, Mondon S, Barrio P, Andreu M, Raich A, Bernabeu J, Vilaplana J, Roca X, Bautista P, Guydish J, Martinez C; group of clinicians involved in the recruitment of the study. Tobacco cessation among smokers under substance use treatment for alcohol and/or cannabis: study protocol and pilot study. Addict Sci Clin Pract. 2022 Nov 30;17(1):66. doi: 10.1186/s13722-022-00348-9. PMID 36451226